CLINICAL TRIAL: NCT01508091
Title: Calorie Restriction Retards the Aging Process by Inducing Sirtuins and Uncoupling Protein 3, Thereby Reducing the Production of Reactive Oxygen Species.
Brief Title: Calorie Restriction Retards the Aging Process
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, MARIA PIA DE LA MAZA, MD, University of Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FONDECYT 1110035
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
Keywords: Obesity; ageing
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calorie restricted (Experimental): 25 % calorie restriction respect measured total energy expenditure, using a Mediterranean diet
  Interventions: Behavioral: energy restricted mediterranean-type diet; Behavioral: 25 % calorie restriction

INTERVENTIONS:
Behavioral: energy restricted mediterranean-type diet — Prescription of diet 25 % lower than actual total energy expenditure in overweight or moderately obese premenopausal women
  Other Names: Calorie restriction; Energy restriction; Mediterranean diet
Behavioral: 25 % calorie restriction — 25 % calorie restriction respect total energy expenditure

SUMMARY:
Calorie restriction is the only experimental manipulation that prolongs longevity in experimental animals. The life prolonging effects of calorie restriction are related to a lower incidence of tumors and less inflammation, but more importantly, a lower generation of reactive oxygen species (ROS). This effect is related to the overexpression of two groups of enzymes. One is a group of (NAD+)-dependent deacetylases called sirtuins whose main actions are to increase free fatty acid flow from adipose tissue, improve insulin secretion and promote mitochondrial biogenesis in muscle. The other group corresponds to uncoupling proteins (UCP), specially UCP 3 that reduces the mitochondrial production of ROS. On the other hand, an effect of calorie restriction that is always reported, is a decrease in resting energy expenditure. A reduction in the activity of UCP1 in brown adipose tissue could be a mechanisms to explain this effect. However sirtuins apparently increase the expression of UCP1.Recently PET CT scans have emerged as a non invasive methodology to recognize brown adipose tissue activity and indirectly, UCP1 activity. Also measurement of telomere length in peripheral blood mononuclear cells has consolidated as a good marker of aging. Two possible models of calorie restriction can be studied in humans. One is a retrospective model in which adults are separated in those that have maintained a stable weight during adulthood in a manner analogous to the weight clamp model of calorie restriction in non human primates. This model is only reliable if there are objective records of the weight that the studied subjects had 20 or more years ago. In the retrospective part of this project the investigators propose to study adults whose weight was recorded previously. The investigators pretend to compare telomere length and expression of SIRT1 and 6 in PBMC, plasma 8 isoprostanes and carotid intima media thickness between weight maintainers and weight gainers. The investigators hypothesis is that weight maintainers will have a better aging profile than weight gainers. In the prospective part of the project the investigators will study a human model of calorie restriction prescribing a 25% reduction in calorie intake during 3 months and comparing groups according to weight loss. At baseline and the end of the study period, UCP3 and SIRT1 expression in muscle biopsies, SIRT1 and 6 expression in PBMC and brown adipose activity, assessed by 18fluorodeoxyglucose uptake using PET/CT will measured. The investigators hypothesis is that individuals subjected to calorie restriction will experience an increase in the expression of UCP3, SIRT1 and SIRT6 and a reduction in brown adipose tissue activity. Simultaneously, these subjects will experience a reduction in oxidative stress markers in muscle and plasma.

DETAILED DESCRIPTION:
HYPOTHESIS: Calorie restriction delays the ageing process and thus telomere erosion, due to a reduction of oxidative stress, via expression modulation of uncoupling proteins and sirtuins.

RETROSPECTIVE STUDY:

Approximately 1000 adults aged 40 to 55 years, that had participated in nutritional assessments studies during which their body weight was recorded, and had a body mass index (BMI) of less than 30 kg/m2 at that time will be considered eligible. Other sources of subject recruitment will be health records from armed forces personnel and our institutional data base. Those that accept and sign a written informed consent, will be subjected to:

1. A complete clinical history, recording past and present diseases, medication use, history of smoking, drinking and illicit drug use.
2. A dietary questionnaire to assess nutrient intake
3. A complete clinical examination including the measurement of body weight, height, blood pressure.
4. A physical activity questionnaire previously validated by us 1
5. Measurement of body composition by DEXA
6. Withdrawal of a 10 hours fasting blood sample of 30 ml to measure

   * Packed red cell volume, blood glucose, creatinine, serum lipids, TSH, thyroid hormones and insulin
   * Telomere length in peripheral blood mononuclear cells (PBMC)
   * Sirt1 and 6 gene expression in PBMC.
   * Plasma 8- isoprostanes
7. Measurement of carotid intima media thickness by ultrasound, performed by a trained professional using previously reported protocols.

Once evaluated, subjects will be classified as:

1. Weight maintainers if their actual weight is, at the most within 10% of the weight recorded at least 10 years before
2. Weight gainers, if their actual weight is over 20% of the weight previously recorded

The following will be excluded from further analysis:

1. Subjects with a history of chronic debilitating diseases such as renal failure, cancer, autoimmune diseases,hypothyroidism, diabetes mellitus or AIDS.
2. Subjects engaged in extremely high physical activity (more than 10 hour per week of sports or work requiring extreme physical activity such as shoveling or hard manual work.
3. Subjects with a history of drug abuse or alcoholism
4. Subjects using anorexigenic or anabolic drugs, or chronic users of non steroidal anti-inflammatory drugs.
5. Subjects smoking more than 5 cigarettes per day (91 packs per year)
6. Overly malnourished subjects, defined as a body mass index below 18 kg/m2.

PROSPECTIVE STUDY:

Main objective:

To study the effects of a three month period of calorie restriction in normal volunteers on the expression of expression of SIRT1 and UCP3 in muscle, SIRT6 in PBMC, brown adipose tissue activity and the accumulation of markers of oxidative damage.

Specific goals:

1. To develop a prospective model of calorie restriction in normal human volunteers.
2. To study changes associated with calorie restriction on:

   * Serum markers of inflammation and free fatty acids during fasting.
   * The uptake of 18fluorodexoyglucose by brown adipose tissue measured by PET-CT
   * The expression of mRNA of UCP3 and SIRT1 in muscle biopsies.
   * The expression of mRNA for SIRT1 and 6 in muscle and peripheral blood mononuclear cells
   * The accumulation of 4 hydroxynonenal and 8 hydroxyguanosine in muscle, as markers of oxidative damage
   * The production of ROS by peripheral neutrophils as an overall measure of the capacity to generate free radicals
   * Insulin sensitivity, measured using formula derived from glucose tolerance. METHODOLOGY Premenopausal women, aged 25 to 40 years, with a BMI between 27 and 32 kg/m2, interested in losing weight, will be studied. Inclusion criteria will be: complete high school, stable weight (± 2 kg) in the last six months, and absence of diabetes, medication intake that could influence energy expenditure such as beta blockers (except oral contraceptives) and lack of engagement in competitive or exhausting physical activities. Women will be required to use an effective contraceptive method, and a pregnancy test will be performed every month while the study lasts.

After signing an informed consent form, total energy expenditure will be measured through calorimetry and actigraphy or doubly labeled water. Subjects will be considered to be in energy balance, taking into account that weight is stable (the lack of weight change will be assessed during the two weeks required for inclusion studies). Therefore, it can be assured that energy intake at that moment is equal to total energy expenditure .

Afterwards, subjects subjected to a 25% restriction of their measured total energy expenditure (this level of restriction has been well tolerated by volunteers, even during one year). Restriction will be balanced, using a mediterranean type diet, maintaining a proportion of 50% carbohydrates, 25-30% of lipids, 25% of proteins and a provision of 100% of micronutrient requirements. Patients will attend to dietician reinforcement every week. To ease the restriction period, one extra meal will be allowed once a week. According to weight change, volunteers will be considered as energy restricted (group 1) is they loose at least 3 kg or 5 % weight during the study period. Instead those subjects that do not reach these goals will be considered as the control group (Group 2).

The intervention will last three months and will be carried out during a period in which temperature remains relatively stable and is lower, in Santiago Chile, to avoid an effect of climate on brown adipose tissue activity. The ideal will be between May and August. Both groups will be evaluated on a weekly basis by a nutritionist to assess compliance with the diet, reinforce indications and be weighed. Subjects will receive a monthly monetary remuneration in order to permit the purchase of specific foods and brands prescribed. Each subject will be educated about healthy dietary and physical activity lifestyle. Eventual changes in physical activity which will be ascertained using portable actigraphs (Actiheart®).

Apart from weight change, volunteers will be considered as calorie restricted if triglyceride levels decrease at least 15% and T3 levels are reduced by at least 8 ng/dl.

At baseline, and the end of the three month intervention period in which controls should be in zero energy balance and adherent subjects in negative energy balance, the following determinations will be carried out:

1. Measurement of routine clinical laboratory parameters to discard concomitant diseases.
2. Measurement of fasting serum free fatty acids.
3. Measurement of ultrasensitive C reactive protein and carboxymethyllisine (CML) as an inflammation marker and glycotoxin respectively, using commercial ELISA kits.
4. Measurement of triglyceride and T3 levels to assess compliance with calorie restriction.
5. Glucose tolerance curve to measure glucose and insulin and calculate insulin sensitivity using Matsuda formula
6. Measurement of oxidative burst of peripheral neutrophils by Fluorescence Activated Cell Sorting (FACS) as an expression of ROS production capacity of the organism
7. Measurement of SIRT1 and 6 gene expression in PBMC by RT-PCR according to the technique reported by Crujeiras et al
8. PET CT to measure 18fluorodeoxyglucose uptake by supraclavicular fat in thermoneutral conditions and after immersing one foot in water at 8°C during five minutes, according to Virtanen et al.
9. Vastus lateralis muscle biopsy, performed by a physician using a Bard needle using a technique previously reported buy our group (this is a safe and simple procedure but the biopsy sample obtained is small, therefore the analyses that can be performed are limited), to measure:

   * mRNA for UCP3 by RT-PCR , using the technique reported by Millet et al in biopsies obtained in a similar way in humans.
   * mRNA for SIRT1 by RT-PCR using the technique reported by Heilbronn et al.
   * Immunohistochemical expression of 8 hydroxyguanosine and 4 hydroxynonenal as oxidation markers, using methods previously reported by us.
10. Body composition measurement by double energy X ray absorptiometry (DEXA).
11. Resting energy expenditure measurement in and open-circuit indirect calorimeter (model 2900, Sensor Medics Corp., Yerba Linda, CA, USA).
12. Actigraphy using Actiheart actigraphs to assess eventual changes in spontaneous physical activity induced by calorie restriction.

Telomere length will not be measured in the prospective protocol, considering that not changes will be detected in the short study period.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese premenopausal women aged 25 - 40 years

Exclusion Criteria:

* diabetes,
* chronic diseases,
* extreme physical exercise,
* drugs affecting energy expenditure

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
UCP3 mRNA expression in vastus lateralis after energy restriction | 3 months
  The main outcome measure will be UCP3 mRNA expression in vastus lateralis, which will be measured before and after the 3 month intervention period. This enzyme is the last link in the chain of events that occur after calorie restriction. Millet et al reported a value for UCP3 mRNA of 15 ± 1.5 amol/ìg total RNA in 18 subjects. Expecting a 60% increase over baseline in the expression of the enzyme, 17 subjects per group are required to obtain results with an á of 0.05 and a power of 0.8. Considering attrition rates, we must study 24 subjects per group.

SECONDARY OUTCOMES:
Brown adipose tissue (BAT) activity, indicating UCP1 expression after calorie restriction | 3 months
  Active BAT and its activation with cold exposure in humans, was demonstrated measuring 18 fluorodeoxyglucose uptake using PET-CT and colocalized the areas of 18F-FDG uptake to the expression of UCP1 thus for practical purposes it is a non invasive and reliable method to detect the presence of the tissue and the activity of UPC1, whic is downregulated by energy restriction.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile